CLINICAL TRIAL: NCT04120818
Title: Expression Profile of Inflammatory Cytokines in Congenital Cataract After Lensectomy and Anterior Vitrectomy
Brief Title: Inflammatory Cytokines in Congenital Cataract After Lensectomy and Anterior Vitrectomy
Status: Completed | Type: Observational
Sponsor: yin ying zhao (Other)
Responsible Party: Sponsor-Investigator, yin ying zhao, Clinical professor, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: yyzhao
Record Dates: First submitted 2019-06-19; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Congenital Cataract
Keywords: inflammatory cytokines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIOL group: aphakic children diagnosed with congenital cataract who underwent secondary IOL implantation
  Interventions: Procedure: secondary IOL implantation
- PIOL group: children with congenital cataract who underwent lensectomy and anterior vitrectomy and primary IOL implantation
  Interventions: Procedure: primary IOL implantation

INTERVENTIONS:
Procedure: secondary IOL implantation — reopened the fibrotic, closed capsular bag and achieve IOL placement
  Groups: SIOL group
Procedure: primary IOL implantation — lensectomy and anterior vitrectomy and primary IOL implantation
  Groups: PIOL group

SUMMARY:
In this prospective study , a cohort of 58 eyes with congenital cataract from Wenzhou medical university was erolled.33 eyes with congenital cataract was after lensectomy and anterior vitrectomy as post-surger group, 26 eyes without cataract surgery as control group. The cytokines of MCP-1, VEGF, IL-1, IFN-γ, IL-1r,IL-4,IL-17, IL-2,IL-5,G-CSF,IL-12, IL-15 was evaluated

DETAILED DESCRIPTION:
Secondary IOL implantation in aphika children and lensectomy and anterior vitrectomy and primary IOL implantation in children with congenital cataract were both performed by the same surgeon(Z.Y.E) and videos were collected to review the capsular reconstruction condition and lens implantation position.

Aqueous humor (100-200 μl) was aspirated from each patient before the surgery. The research was to evaluate the relationship between the cytokine profile in aqueous humor and the state of capsule after Lensectomy and Anterior Vitrectomy.Aqueous humor was obtained , Human Magnetic Luminex Screening Assay was used to determine the aqueous humor levels of cytokines.

ELIGIBILITY:
Inclusion Criteria: aphakic children diagnosed with congenital cataract who underwent secondary IOL implantation and children with congenital cataract who underwent lensectomy and anterior vitrectomy and primary IOL implantation

Exclusion Criteria:patients with mild cataracts do not require surgery

-

Ages: 10 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: congenital cataract age from 10 months to 72 months who underwent cataract surgery or aphakic children age from 15 months to 72 months who underwent secondary IOL implantation
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2017-02-12 (Actual); Study Completion 2017-02-12 (Actual)

PRIMARY OUTCOMES:
inflammatory cytokines | before the surgery of secondary IOL implantation
  investigate inflammatory microenvironment changes in the aqueous of children after surgery.aqueous humor levels of cytokines, chemokines and growth factors including TGFβ2, TNF-α, IL-6, IP10, IL-10, MCP-1, VEGF, IL-1, IFN-γ, IL-1r,IL-4,IL-17, IL-2,IL-5,G-CSF,IL-12, IL-15.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Eye Hosptial of Wenzhou Medical College, Wenzhou, Zhejiang
  - Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang